CLINICAL TRIAL: NCT02632396
Title: A Phase I/II Study of MLN9708 as Post-Transplant Maintenance for Patients With Mantle Cell Lymphoma Undergoing Autologous Stem Cell Transplant in First Remission
Brief Title: Ixazomib & Rituximab After Stem Cell Transplant in Treating Patients With Mantle Cell Lymphoma in Remission
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Emory University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jonathon Cohen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076016; NCI-2015-01943 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); X16058 (Other: Millenium Pharmaceuticals, Inc.); Winship2839-15 (Other: Emory University/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ixazomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ixazomib, rituximab) (Experimental): Beginning between 70-180 days after stem cell transplant, patients receive ixazomib PO on days 1, 8, and 15, and rituximab IV (or SC after first dose if deemed appropriate) on day 1 of courses 1, 3, 5, 7, and 9. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Biological: Rituximab

INTERVENTIONS:
Drug: Ixazomib — Given PO
  Other Names: Ninlaro; MLN9708; Ixazomib Citrate
Biological: Rituximab — Given IV
  Other Names: Rituxan; MabThera; Chimeric Anti-CD20 Antibody

SUMMARY:
This phase I/II trial studies the side effects and best dose of ixazomib citrate (ixazomib) when given together with rituximab and to see how well they work after stem cell transplant in treating patients with mantle cell lymphoma that are no longer showing signs or symptoms of cancer. Ixazomib may stop the growth of cancer cell by blocking enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, may interfere with the ability of cancer cells to grow and spread. Giving ixazomib together with rituximab after transplant may help prevent the cancer from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose and assess the safety of ixazomib when administered as post-transplant maintenance in mantle cell lymphoma and to evaluate the safety of rituximab in combination with the recommended phase II dose (RP2D) of ixazomib. (Phase I)

II. To assess preliminary evidence of efficacy of ixazomib in combination with rituximab when administered as post-transplant maintenance in mantle cell lymphoma. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate for preliminary evidence of efficacy of ixazomib (+/- rituximab) maintenance therapy in patients with mantle cell lymphoma undergoing autologous stem cell transplant in first partial or complete remission. (Phase I)

II. To evaluate for preliminary evidence of efficacy of ixazomib (+/- rituximab) maintenance therapy in patients with mantle cell lymphoma who have a complex karyotype and other high-risk cytogenetic or clinical markers. (Phase I)

III. To evaluate toxicities associated with prolonged administration of ixazomib maintenance therapy in patients with mantle cell lymphoma (MCL). (Phase I)

IV. To evaluate the rate of minimal residual disease (MRD) in patients who have completed an autologous transplant for mantle cell lymphoma and to assess the impact of MRD on outcomes for patients receiving maintenance therapy. (Phase I)

V. To evaluate efficacy of ixazomib with rituximab maintenance therapy in patients with MCL who undergo autologous stem cell transplantation in first remission who have a complex karyotype and/or additional high risk cytogenetic or clinical features at diagnosis. (Phase II)

VI. To further evaluate safety and toxicity of prolonged administration of ixazomib. (Phase II)

VII. To evaluate long-term disease-related and survival outcomes for patients with MCL who receive post-transplant maintenance therapy with ixazomib with rituximab. (Phase II)

VIII. To evaluate the rate of minimal residual disease (MRD) in patients who have completed an autologous transplant for mantle cell lymphoma and to assess the impact of MRD on outcomes for patients receiving maintenance therapy. (Phase II)

TERTIARY OBJECTIVES:

I. To evaluate the prognostic value of pre-transplant positron emission tomography (PET)/computed tomography (CT) in mantle cell lymphoma.

II. To evaluate the ability of the single nucleotide polymorphism (SNP) array to identify high-risk cytogenetic features in patients with MCL.

III. To evaluate the impact of ixazomib maintenance (+/- rituximab) on immunoglobulin levels for patients completing autologous stem cell transplantation for mantle cell lymphoma.

OUTLINE: This is a phase I, dose-escalation study of ixazomib followed by a phase II study.

Beginning between 70-180 days after stem cell transplant, patients receive ixazomib orally (PO) on days 1, 8, and 15, and rituximab intravenously (IV) (or subcutaneously [SC] after first dose if deemed appropriate) on day 1 of courses 1, 3, 5, 7, and 9. Treatment repeats every 28 days for up to 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).
* Patients must have a diagnosis of mantle cell lymphoma confirmed at diagnosis by one of the following:

  * t(11;14) detected by fluorescence in situ hybridization (FISH), conventional cytogenetics, or other molecular evaluation
  * Expression of cyclin D1 confirmed by immunohistochemistry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Patients must have completed an autologous stem cell transplant after their first course of treatment; patients who have relapsed or progressed at any time prior to transplant are not eligible.
* Patients must not have experienced confirmed progressive disease since the time of their transplant.
* Absolute neutrophil count (ANC) ≥ 1,000/mm³ and platelet count ≥ 75,000/mm³. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment. Patients may receive growth factor support prior to initiating therapy but must remain off of growth factor for at least 7 days before starting therapy and must meet eligibility on cycle 1, day 1. Patients who complete the consent process but do not meet hematologic eligibility within 30 days may be re-consented and enrolled on study if they ultimately do meet eligibility requirements before day +180. No patients may initiate therapy after day +180 and they must meet all remaining eligibility criteria.
* Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN) except for previously documented Gilbert's disease, defined as a mild unconjugated hyperbilirubinemia with no other identifiable cause and bilirubin values < 6 mg/dL; patients with hyperbilirubinemia secondary to presumed Gilbert's disease who are being considered for enrollment in the study MUST have a fractionated bilirubin included in their screening labs when determining eligibility.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
* Calculated creatinine clearance ≥ 30 mL/min using Cockcroft-Gault formula.
* Note: Patients are expected to initiate therapy as close to day +100 as possible. No patient may initiate therapy before day +70 and initiation of therapy beyond day +130 is allowed ONLY for patients who meet all eligibility criteria except for hematologic parameters, in which case patients may be delayed until their hematologic laboratories meet criteria but no later than day +180. Regardless of the time of therapy initiation, patients must meet all eligibility criteria and must have completed all consent documentation and screening procedures within the specified window.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Failure to have fully recovered (ie, ≤ grade 1 toxicity) from the reversible effects of prior chemotherapy, except for laboratory abnormalities which are addressed above.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib.
* Central nervous system involvement with lymphoma at any time in the patient's history; intrathecal prophylaxis during induction is allowed as long as active disease has not been identified.
* Infection requiring intravenous antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months; patients experiencing an isolated cardiac complication at the time of transplant who have been evaluated by cardiology and remained stable for at least 60 days are eligible.
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong cytochrome P450, family 3, subfamily A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's wort.
* Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive. Patients who have previously tested positive for hepatitis B core antibody may be eligible if they are confirmed to NOT have active disease and are on appropriate anti-viral therapy. No additional hepatitis or HIV testing is required for patients who have been evaluated during their induction and/or pre-transplant work-up and have had no clinical evidence of HIV, hepatitis B or hepatitis C since their last evaluation.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent. Patients with a prior reaction to rituximab are permitted if the investigator feels that this reaction is manageable with standard supportive care measures and would otherwise be comfortable administering rituximab outside of the clinical trial setting.
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing; patients with known GI involvement with mantle cell lymphoma who have no clinical evidence of active disease at the time of enrollment are eligible.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease; patients with non-melanoma skin cancer, carcinoma in situ of any type, or low risk cervical cancer are not excluded if they have undergone complete resection and are deemed free of disease by their treating physician; patients with low risk prostate cancer who are under observation are eligible if their urologist or oncologist does not expect them to require therapy within 1 year.
* Patient has ≥ grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period.
* Receipt of therapy on a clinical trial, including investigational and non-investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial; participation on non-therapeutic clinical studies is allowed, and patients who participated on a clinical trial for induction and/or transplant but who have completed the prescribed therapy course for that study and have been off therapy for at least 30 days are eligible.
* Prior exposure to ixazomib; however, prior bortezomib exposure is allowed.
* Patients with any history of relapsed/refractory disease, or who have progressed at any time since beginning induction therapy are not eligible; patients who have evidence of residual disease by FISH, cytogenetics, SNP array, or flow cytometry without any measurable nodal disease or morphologic evidence of disease in the bone marrow or peripheral blood are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of ixazomib, defined as the dose where 1 or fewer of 6 treated patients experience a dose limiting toxicity graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 (Phase I) | 28 days
Progression-free survival (PFS), defined as the percentage of patients who have received at least one dose of study therapy who are alive and free of disease progression or relapse at 1-year post autologous stem cell transplant (Phase II) | 1 year
  Determined using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Conversion rate from MRD positive to MRD negative during therapy (Phase I & II) | Up to 10 months (10 courses of treatment)
Incidence of adverse events graded according to CTCAE version 4.03 (Phase I & II) | Up to 30 days after administration of the last dose of study treatment
  Adverse events will be tabulated across all patients who received any treatment with a focus on severe (grade 3-5) adverse events and toxicities as well as commonly encountered lower grade adverse events. All adverse events will be reported in tabular form, and as, possible, identification of adverse events possibly, probably, or definitely related to study therapy will be noted.
Median OS (Phase II) | Up to 2 years
  The relationship between cytogenetic variables and OS will be explored using the Kaplan-Meier method.
Median PFS (Phase II) | Up to 2 years
  The relationship between cytogenetic variables and PFS will be explored using the Kaplan-Meier method.
Overall survival (OS) (Phase II) | 1 year
  The relationship between cytogenetic variables and OS will be explored using the Kaplan-Meier method.
PFS for all patients and for those patients with a complex karyotype and other high-risk clinical or cytogenetic features (Phase I) | 1 year
  The relationship between cytogenetic variables and PFS will be explored using the Kaplan-Meier method.
PFS for patients with a complex karyotype and other high risk clinical or cytogenetic features (Phase II) | 1 year
  The relationship between cytogenetic variables and PFS will be explored using the Kaplan-Meier method.
Rate of MRD positivity (Phase I & II) | Baseline
Rate of patients maintaining MRD negativity from study entry to completion of therapy (Phase I & II) | Up to 10 months (10 courses of treatment)

OTHER OUTCOMES:
Median OS for patients who have a pre-transplant PET/CT (Phase II) | Up to 2 years
  The relationship between a pre-transplant PET/CT and outcomes with respect to PFS will be explored for those patients who have available images from prior to transplant.
Median PFS for patients who have a pre-transplant PET/CT (Phase II) | Up to 2 years
  The relationship between a pre-transplant PET/CT and outcomes with respect to PFS will be explored for those patients who have available images from prior to transplant.
PFS for patients who have a pre-transplant PET/CT (Phase II) | 1 year
  The relationship between a pre-transplant PET/CT and outcomes with respect to PFS will be explored for those patients who have available images from prior to transplant.
Recurrent abnormalities identified by SNP array (Phase II) | Up to 2 years
  All patients with available tissue or bone marrow samples will complete a cytogenetic evaluation including FISH for t(11;14) and del(17p) as well as conventional karyotyping and SNP array. Relationships between these variables and response to maintenance therapy will be explored. The relationship between cytogenetic variables and PFS and OS will be explored using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Cohen, MD, MS, Principal Investigator — Emory University/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Romancik JT, Chen Z, Allen PB, Waller EK, Valla K, Colbert A, Rosand C, Palmer AF, Flowers CR, Cohen JB. Ixazomib With or Without Rituximab Following Maintenance Autologous Stem Cell Transplant in Mantle Cell Lymphoma: A Single-Center Phase I Trial. Clin Lymphoma Myeloma Leuk. 2022 Dec;22(12):e1084-e1091. doi: 10.1016/j.clml.2022.08.013. Epub 2022 Aug 24. PMID 36180329

DOCUMENTS (1):
  • Informed Consent Form (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT02632396/ICF_000.pdf